CLINICAL TRIAL: NCT06840652
Title: Safety and Efficacy Assessment of Baclofen for Alcohol Withdrawal in Patients With Chronic Liver Disease and Active Alcohol Consumption
Brief Title: Safety & Efficacy of Baclofen for Alcohol Withdrawal in Chronic Liver Disease With Active Alcohol Consumption
Acronym: BAWIC
Status: Enrolling by invitation | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Jordi Sanchez-Delgado, Head of the Hepatology Hospitalization Unit, Corporacion Parc Tauli
Other Study IDs: 2023/5106; 2023/5106 (Other: Consorci Corporació Sanitària Parc Taulí)
Record Dates: First submitted 2025-01-11; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Alcoholic Cirrhosis; Alcohol Abstinence; Alcohol Withdrawal; Medication Toxicity; Medication Adherence
Keywords: alcohol withdrawal; baclofen; alcoholic cirrhosis; alcohol abstinence
MeSH Terms: conditions — Liver Cirrhosis, Alcoholic; Alcohol Abstinence; Drug-Related Side Effects and Adverse Reactions; Medication Adherence | interventions — Baclofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with alcohol-related cirrhosis who persist in active alcohol consumption.: Patients with alcohol-related cirrhosis with active alcohol consumption and are being monitored in outpatient hepatology clinics. Baclofen treatment will be prescribed by hepatologists and/or psychiatrists and all patients will be referred for follow-up in outpatient addiction clinics.
  Interventions: Drug: Baclofen

INTERVENTIONS:
Drug: Baclofen — Safety and effectiveness of baclofen as a treatment for alcohol withdrawal in patients with chronic liver disease. The investigators will administer baclofen in increasing doses up to a maximum dose of 10 mg every 8 hours, evaluating the drug's tolerance and its effectiveness in achieving alcohol abstinence. Baclofen will be administered during the patient's hospitalization for decompensation of their liver disease, in patients followed up as outpatients in hepatology clinics, and in those managed as outpatients by psychiatrists specializing in addiction

SUMMARY:
This study examines the safety and effectiveness of baclofen as a treatment for alcohol withdrawal in patients with chronic liver disease who continue drinking. It aims to evaluate baclofen's ability to promote alcohol abstinence or reduction while monitoring adverse effects. Secondary outcomes include liver function changes, hospital readmissions, and complications of cirrhosis.

Alcohol consumption worsens liver disease prognosis, yet alcohol use disorder (AUD) often goes untreated. Baclofen, which is safe for patients with liver impairment, is recommended as a first-line treatment for AUD in chronic liver disease. This prospective study collects data from patients treated with baclofen at Parc Taulí Hospital, analyzing outcomes at three and six months to assess abstinence, alcohol reduction, and adverse effects.

DETAILED DESCRIPTION:
The medical management of alcohol use disorder (AUD) requires a multidisciplinary approach, involving psychiatrists, psychologists, and hepatologists. Treatment often combines pharmacotherapy with psychosocial interventions to achieve and maintain abstinence. Over the years, various anti-craving medications have been used. Due to its renal metabolism, rather than hepatic, baclofen is considered safe for individuals with chronic liver disease and is currently the first-line pharmacological agent for patients with AUD and secondary liver disease.

Despite clinical guidelines recommending baclofen as the preferred medication to reduce alcohol consumption in patients with chronic liver disease, its use remains limited. Moreover, no published data or communications exist regarding its application in the investigators specific context.

The primary objectives of this study are to assess the rate of abstinence maintenance, evaluate the reported reduction in alcohol consumption, and assess the safety of baclofen as a treatment for alcohol abstinence.

The secondary objectives include evaluating changes in liver function related to alcohol abstinence or consumption reduction. Liver function will be assessed using the CHILD Score (Child-Turcotte-Pugh, CTP) and the MELD Score (Model for End-Stage Liver Disease), both of which are essential tools for predicting prognosis in patients with cirrhosis.

Treatment initiation may occur across various hospital settings, including inpatient units during hospitalizations, outpatient hepatology services, and psychiatric services.

The investigators will evaluate the efficacy and safety of baclofen through regular follow-ups with patients who initiate treatment. Data collection methods will include patient interviews, self-reported abstinence, blood tests to assess liver function, and baseline information on active drinking behavior. Follow-up will be conducted over a period of six months

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic liver disease at any stage
* Active alcohol consumption
* Use of baclofen for the treatment of alcohol dependence.

Exclusion Criteria:

* Severe psychiatric illness requiring other psychotropic pharmacological treatments
* Organic or functional renal insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A single-center retrospective study of patients with alcohol-related chronic liver disease (alcoholic liver disease and cirrhosis) who receive baclofen as treatment for alcohol dependence.
  The treatments have been initiated from different hospital settings: 1) Inpatient units during hospitalization for complications of liver disease, 2) Outpatient care setting provided by hepatologists 3) Patiens with cirrhosis in emergency care setting and 4) Outpatient care setting provided by psychiatrists.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who achieve abstinence | During 6 months
  The investigators will report, through clinical interviews, the percentage of patients who have stopped drinking
Rate of patients who reduce alcohol consumption | During 6 months
  The investigators will report, through clinical interviews, the percentage of patients who have reduced alcohol consumption

SECONDARY OUTCOMES:
Rate of patients discontinuing treatment due to side effects | During 6 months
  The investigators will report, through clinical interviews, the tolerance and side effects of the baclofen
CHILD and MELD score improvement if abstinence is achieve | During 6 months
  The investigators will evaluate the improvement in liver function in relation to abstinence measured by CHILD and MELD scores.
  The Child-Pugh classification assesses the prognosis of cirrhosis, using five parameters: Total Bilirubin (mg/dL), Serum Albumin (g/dL), Prothrombin Time (PT) or INR, Ascites, and Hepatic Encephalopathy. Each is scored from 1 to 3 points, with higher scores indicating worse liver function. The total score categorizes patients into: Class A (5-6 points) - mild disease with good liver function, Class B (7-9 points) - moderate severity, and Class C (10-15 points) - severe liver dysfunction with poor prognosis.
  The MELD score (Model for End-Stage Liver Disease) predicts short-term mortality using Serum Bilirubin, Serum Creatinine, and INR. Low MELD (<15) suggests low mortality risk, High MELD (≥15) indicates significant dysfunction, and Very High MELD (≥30) reflects critical liver failure, prioritizing for transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Sánchez Delgado, MD. PhD, Principal Investigator — Consorci Corporació Sanitària Parc Taulí
Locations (1):
- Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share our preliminary results with other interested researchers in case they are interested in conducting a multicenter study
Supporting Information: SAP
Time Frame: The supporting information will be available in january'26 till january'27
Access Criteria: Other investigators will be able to access to this information by contacting by email with the principal investigator

REFERENCES:
- [Background] Agabio R, Sinclair JM, Addolorato G, Aubin HJ, Beraha EM, Caputo F, Chick JD, de La Selle P, Franchitto N, Garbutt JC, Haber PS, Heydtmann M, Jaury P, Lingford-Hughes AR, Morley KC, Muller CA, Owens L, Pastor A, Paterson LM, Pelissier F, Rolland B, Stafford A, Thompson A, van den Brink W, de Beaurepaire R, Leggio L. Baclofen for the treatment of alcohol use disorder: the Cagliari Statement. Lancet Psychiatry. 2018 Dec;5(12):957-960. doi: 10.1016/S2215-0366(18)30303-1. Epub 2018 Nov 6. No abstract available. PMID 30413394
- [Background] Duan F, Zhai H, Liu C, Chang C, Song S, Li J, Cheng J, Yang S. Systematic review and meta-analysis: Efficacy and safety of baclofen in patients with alcohol use disorder co-morbid liver diseases. J Psychiatr Res. 2023 Aug;164:477-484. doi: 10.1016/j.jpsychires.2023.06.042. Epub 2023 Jun 30. PMID 37441998
- [Background] Mekonen T, Chan GCK, Connor J, Hall W, Hides L, Leung J. Treatment rates for alcohol use disorders: a systematic review and meta-analysis. Addiction. 2021 Oct;116(10):2617-2634. doi: 10.1111/add.15357. Epub 2021 Jan 12. PMID 33245581
- [Background] Glantz MD, Bharat C, Degenhardt L, Sampson NA, Scott KM, Lim CCW, Al-Hamzawi A, Alonso J, Andrade LH, Cardoso G, De Girolamo G, Gureje O, He Y, Hinkov H, Karam EG, Karam G, Kovess-Masfety V, Lasebikan V, Lee S, Levinson D, McGrath J, Medina-Mora ME, Mihaescu-Pintia C, Mneimneh Z, Moskalewicz J, Navarro-Mateu F, Posada-Villa J, Rapsey C, Stagnaro JC, Tachimori H, Ten Have M, Tintle N, Torres Y, Williams DR, Ziv Y, Kessler RC; WHO World Mental Health Survey Collaborators. The epidemiology of alcohol use disorders cross-nationally: Findings from the World Mental Health Surveys. Addict Behav. 2020 Mar;102:106128. doi: 10.1016/j.addbeh.2019.106128. Epub 2019 Sep 16. PMID 31865172
- [Result] Rehm J, Mathers C, Popova S, Thavorncharoensap M, Teerawattananon Y, Patra J. Global burden of disease and injury and economic cost attributable to alcohol use and alcohol-use disorders. Lancet. 2009 Jun 27;373(9682):2223-33. doi: 10.1016/S0140-6736(09)60746-7. PMID 19560604
- [Result] GBD 2016 Alcohol Collaborators. Alcohol use and burden for 195 countries and territories, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet. 2018 Sep 22;392(10152):1015-1035. doi: 10.1016/S0140-6736(18)31310-2. Epub 2018 Aug 23. PMID 30146330